CLINICAL TRIAL: NCT02646592
Title: Effect of a Bolus of 10 µg/kg of Alfentanil on the Pupillary Pain Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pr Isabelle CONSTANT (Other)
Responsible Party: Sponsor-Investigator, Pr Isabelle CONSTANT, Professor, Hôpital Armand Trousseau
Organization: Hôpital Armand Trousseau (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PPI Alfentanil
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Pain; Anesthesia
MeSH Terms: conditions — Pain | interventions — Alfentanil; Sevoflurane; Propofol

ARMS (1):
- alfentanil (Experimental): Children under general anesthesia for elective surgery. Induction with sevoflurane or propofol according to the preference of the patient.
  Maintenance with sevoflurane. 5 minutes before skin incision, first assessment of the pupillary pain index. Then injection of 10 µg/kg of alfentanil. After 5 minutes second assessment of pupillary pain index. End of study period, beginning of surgery.
  Interventions: Drug: Alfentanil; Drug: sevoflurane or propofol

INTERVENTIONS:
Drug: Alfentanil — Bolus of alfentanil 10 µg/kg 5 minutes before skin incision
Drug: sevoflurane or propofol

SUMMARY:
This study aims to assess the Pupillary Pain Index before and after a bolus of alfentanil in children under general anesthesia, before skin incision.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery under general anesthesia
* Written informed consent

Exclusion Criteria:

* Chronic pain
* Preoperative analgesic drug
* Neurologic disease
* Ophtalmic disease

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change between Pupillary Pain Index before and after alfentanil bolus | Five minutes before incision and just before incision. Each measure = 20 seconds
  pupillometry

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Constant, PHD, Study Director — University Hospital Armand Trousseau
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France

REFERENCES:
- [Derived] Sabourdin N, Diarra C, Wolk R, Piat V, Louvet N, Constant I. Pupillary Pain Index Changes After a Standardized Bolus of Alfentanil Under Sevoflurane Anesthesia: First Evaluation of a New Pupillometric Index to Assess the Level of Analgesia During General Anesthesia. Anesth Analg. 2019 Mar;128(3):467-474. doi: 10.1213/ANE.0000000000003681. PMID 30198934